CLINICAL TRIAL: NCT00605163
Title: A Longitudinal Observational Follow-up of the PRECEPT Study Cohort
Acronym: PostCEPT
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: The Parkinson Study Group (Network)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); H. Lundbeck A/S (Industry); Parkinson's Disease Foundation (Other); United States Department of Defense (U.S. Federal Agency)
Responsible Party: Ira Shoulson, MD, Principal Investigator, University of Rochester Clinical Trials Coordination Center
Other Study IDs: U01NS050095_PostCEPT; NINDS 5 U01NS050095-02; U01NS050095 (NIH)
Record Dates: First submitted 2008-01-17; First posted 2008-01-30 (Estimated); Last update posted 2008-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Parkinson Disease
Keywords: Parkinson disease, observational, longitudinal
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort
Biospecimen Retention: Samples With DNA — Whole blood
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to longitudinally follow consenting clinical trial participants who participated in PRECEPT (A Randomized, Double Blind, Placebo Controlled, Dose Finding Study to Assess the Efficacy and Safety of CEP 1347 in Patients With Early Parkinson's Disease). The study will assess the clinical and imaging outcomes relevant to the natural history of Parkinson's disease (PD), as well as determine early biomarkers of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the PRECEPT study
* Willing and able to give informed consent

Exclusion Criteria:

* Patients will be excluded from participating in the the study if either of the criteria stated above is not met

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Parkinson disease patients who participated in the PRECEPT clinical trial.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2006-08; Primary Completion 2010-08 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson Disease Rating Scale (UPDRS) and β-CIT SPECT imaging of the dopamine transporter. | Annual, ongoing assessments

SECONDARY OUTCOMES:
University of Pennsylvania Smell Identification Test (UPSIT) | Annual, ongoing assessments

CONTACTS AND LOCATIONS:
Locations (55):
- United States (47):
  - Barrow Neurological Institute, Phoenix, Arizona
  - Sun Health Research Institute, Sun City, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - The Parkinson's & Movement Disorder Institute, Fountain Valley, California
  - University of California Irvine, Irvine, California
  - University of San Diego, La Jolla, California
  - University of Southern California, Los Angeles, California
  - Pacific Neuroscience Medical Group, Oxnard, California
  - University of California Davis, Sacramento, California
  - The Parkinson's Institute, Sunnyvale, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Colorado Neurological Institute, Littleton, Colorado
  - Institute for Neurogenerative Disorders, New Haven, Connecticut
  - Mayo Clinic Jacksonville, Jacksonville, Florida
  - University of South Florida, Tampa, Florida
  - Cleveland Clinic Florida-Weston, Weston, Florida
  - Medical College of Georgia, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kansas Medical Center, Kansas City, Kansas
  - LSU Health Science Center Shreveport, Shreveport, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Boston University, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Minnesota, Minneapolis, Minnesota
  - Creighton University, Omaha, Nebraska
  - UMDNJ Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Albany Medical College, Albany, New York
  - North Shore-LIJ Health System, Manhasset, New York
  - Beth Israel Medical Center, New York, New York
  - Columbia University, New York, New York
  - University of Rochester, Rochester, New York
  - Duke University Medical Center, Durham, North Carolina
  - University of Cincinnati/Cincinnati Children's Hospital, Cincinnati, Ohio
  - Oregon Health & Science University, Portland, Ohio
  - Medical University of Ohio, Toledo, Ohio
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - NeuroHealth Parkinson's Disease Movement Disorders Center, Warwick, Rhode Island
  - University of Tennessee-Memphis, Memphis, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - University of Virginia, Charlottesville, Virginia
- Canada (8):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - London Health Sciences Centre, London, Ontario
  - Ottawa Hospital Civic Site, Ottawa, Ontario
  - Toronto Western Hospital, University Health Network, Toronto, Ontario
  - University of Sherbrooke, Fleurimont, Quebec
  - Hotel-Dieu Hospital-CHUM, Montreal, Quebec
  - Saskatoon Disrict Health Board Royal University Hospital, Saskatoon, Saskatchewan

REFERENCES:
- [Background] Parkinson Study Group PRECEPT Investigators. Mixed lineage kinase inhibitor CEP-1347 fails to delay disability in early Parkinson disease. Neurology. 2007 Oct 9;69(15):1480-90. doi: 10.1212/01.wnl.0000277648.63931.c0. Epub 2007 Sep 19. PMID 17881719
- [Derived] Latourelle JC, Beste MT, Hadzi TC, Miller RE, Oppenheim JN, Valko MP, Wuest DM, Church BW, Khalil IG, Hayete B, Venuto CS. Large-scale identification of clinical and genetic predictors of motor progression in patients with newly diagnosed Parkinson's disease: a longitudinal cohort study and validation. Lancet Neurol. 2017 Nov;16(11):908-916. doi: 10.1016/S1474-4422(17)30328-9. Epub 2017 Sep 25. PMID 28958801
- See also: The Parkinson Study Group (PSG) is a non-profit, cooperative group of Parkinson's disease experts from medical centers in theUnited States and Canada who are dedicated to improving treatment for persons affected by Parkinson's disease. — http://www.Parkinson-Study-Group.org